CLINICAL TRIAL: NCT01904773
Title: A 6-month, Multicenter, Randomized, Safety, Tolerability, Pharmacokinetic, and Preliminary Efficacy Study of AZD5213 in Adolescents With Tourette's Disorder
Brief Title: Safety, Tolerability, Pharmacokinetic, and Efficacy Study of AZD5213 in Adolescents With Tourette's Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D3032C00001
Record Dates: First submitted 2013-07-18; First posted 2013-07-22 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Tourette Syndrome
Keywords: Combined Multiple Motor and Vocal Tic Disorder; Tourette Disorder; Gilles de la Tourette Syndrome; Tourette Disease
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: AZD5213 and placebo
- low dose AZD5213 (Experimental)
  Interventions: Drug: AZD5213 and placebo
- high dose AZD5213 (Experimental)
  Interventions: Drug: AZD5213 and placebo

INTERVENTIONS:
Drug: AZD5213 and placebo — low dose AZD5213 capsules; high dose AZD5213 capsules; placebo capsules

SUMMARY:
This is a two-part, randomized, multi-center, blinded study in adolescents with Tourette's Disorder. There will be an up to 21-day screening period in which subject eligibility will be determined. In Part 1 of the study, the safety, tolerability and pharmacokinetics of AZD5213 will be assessed during a 1- week period.

In Part 2 of the study, the safety, tolerability, and preliminary efficacy of two doses (depending on tolerability in Part 1 of the study) of AZD5213 and placebo will be assessed through six consecutive four-week crossover periods. Each subject will receive both AZD5213 and placebo. A follow-up vist will take place at 14 (±) 7 days following the last dose of study drug.

DETAILED DESCRIPTION:
This is a multicenter, randomized, two-part study of AZD5213 in adolescents (ages 12-17 years) with Tourette's Disorder.

In Part 1 of the study, following an up to 21-day screening period, on Day 1, after baseline procedures are performed, eligible subjects will receive a single, low dose of AZD5213, in-clinic.

After study drug dosing on Day 1, safety and tolerability will be assessed in-clinic, and blood samples will be taken for pharmacokinetic (PK) analysis. On Days 2, 3, 4, 5, 6 and 7 subjects will take study drug, and will be contacted via telephone and adverse events and concomitant medications will be assessed. On Day 8, safety, tolerability, and blood sampling for PK analysis (predose and 2-4 hours post-dose) will be performed in-clinic. Part 2 of the study will consist of six consecutive crossover periods. In Part 2 of the study, each study drug will be administered in two 4-week periods (six treatment periods, total). Each study drug will be received in one of Periods 1-3, and again in one of Periods 4-6. Approximately 24 subjects will receive study drug in Part 1 of this study in order to complete approximately 18 subjects in Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between the ages of ≥ 12 and < 18 years at baseline (Day 1).
2. Meets Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for Tourette's Disorder, as assessed by the Kiddie-SADS (Schedule for Affective Disorders and Schizophrenia)-Present and Lifetime Version (K-SADS-PL) Tic Disorder Supplement and clinical interview.
3. Yale Global Tic Severity Scale (YGTSS) Total Tic Severity Score (TTS) ≥ 20 at Screen and baseline (Day 1).
4. Symptoms of Tourette's Disorder must impair school, occupational, and/or social function.
5. Written informed assent or consent provided by the subject, and written informed consent provided by the parent(s)/guardians(s), as appropriate per the Institutional Review Board/Ethics Committee. 6. Weight ≥ 40 kg at the screening and baseline (Day 1) visits.

7. In the opinion of the investigator, the subject and designated guardian(s) and/or parent(s) must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Prior participation in any AZD5213 study.
2. Acute suicidality as evidenced by answering "yes" for question #4 or question #5 on the Columbia-Suicide Severity Rating Scale (C-SSRS), indicating active suicidal ideation with any intent to act, at Screen or baseline (Day 1).
3. Pregnant or breast-feeding females.
4. History of seizure disorder other than a single childhood febrile seizure.
5. Presence of any psychiatric or neurologic disorder or symptom, if, in the judgment of the investigator, the psychiatric or neurologic disorder or symptom is likely to confound interpretation of drug effect or affect the subject's ability to complete the study. 6. Any clinically important abnormality as determined by the investigator at Screen or baseline (Day 1) in physical or neurologic examination, vital sign, ECG, or clinical laboratory test results that could be detrimental to the subject or could affect the subject's ability to complete the study.

7. History or presence of any clinically important medical condition that, in the judgement of the investigator, is likely to deteriorate, could be detrimental to the subject, or could affect the subject's ability to complete the study.

8. History or presence of a clinically important sleep disorder.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Research Site, Orange, California
  - Research Site, St. Petersburg, Florida
  - Research Site, Summit, New Jersey
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Orem, Utah
  - Research Site, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects between the ages of 12 and 17 with Tourette's Disorder
Pre-assignment Details: There were 29 screening visits for 28 subjects, 1 subject was initially screen failed for exclusion 32 but rescreened and qualified and entered Part 1 of the study(104-4003 rescreened and qualified as 104-4004). Eligible subjects participated in Part 1 and then continued into a randomized 6 period crossover Part 2 of the study
Groups:
- Initial Study: Initial Screen, Part 1: AZD5213 0.5 mg single dose Day 1, AZD5213 2 mg dose Days 6-8
- Part 2 -Sequence BBABBA; Part 2- Sequence BABBAB: B=AZD5213 0.5 mg, A=Placebo (did not tolerate 2.0 mg in Part 1)
- Part 2 - Sequence ABCACB; Part 2- Sequence BACCAB; Part 2- Sequence BCACBA; Part 2 Sequence CABBAC; Part 2- Seqence CBABCA: A=Placebo, B=AZD5213 0.5 mg, C=AZD5213 2.0 mg
- Part 2- Sequence ACBABC: A= Placebo, B=AZD5213 0.5 mg, C=AZD5213 2.0 mg
Period: Screen
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Screen failure | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 - Single Dose- AZD5213 0.5 mg
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 - Multiple Dose AZD5213 2.0 mg
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tolerated 2.0 mg in Part 1 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Did Not Tolerate 2.0 mg in Part 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: First Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 2 | 1 | 2 | 3 | 4 | 4 | 3 | 4
Completed | 0 | 2 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Placebo Washout First Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 2 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Completed | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Condition worsened | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Completed | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Placebo Washout Second Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Completed | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Completed | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Placebo Washout Third Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Completed | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Completed | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Placebo Washout Fourth Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Completed | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fifth Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 3 | 4
Completed | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Placebo Washout Fifth Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 1 | 1 | 2 | 3 | 4 | 3 | 2 | 4
Completed | 0 | 0 | 1 | 2 | 3 | 4 | 3 | 2 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study specific withdrawal criteria | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Sixth Intervention
Arm/Group | Initial Study | Part 2 -Sequence BBABBA | Part 2- Sequence BABBAB | Part 2 - Sequence ABCACB | Part 2- Sequence ACBABC | Part 2- Sequence BACCAB | Part 2- Sequence BCACBA | Part 2 Sequence CABBAC | Part 2- Seqence CBABCA
Started | 0 | 0 | 1 | 2 | 3 | 4 | 3 | 2 | 4
Completed | 0 | 0 | 1 | 2 | 3 | 4 | 3 | 2 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled in Part 1 of the study, 23 of whom continued into Part 2
Groups:
- Overall Study: Part 1 & Part 2
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Adolescent - age 12 to 17
  years | 14.6 (1.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Nicotine use [Number; unit: Participants] — Have ever used nicotine, never, past, present response
  Participants
    Current | 0
    Never | 24
    Past | 0
Tourette's Disorder Duration [Median (Full Range); unit: months] — Tourette's Disorder Duration in months
  months | 75 [29.8 to 159.4]

OUTCOME MEASURES:

1. Primary Outcome: Total Tic Severity Score (Part 2 Only) Crossover Analysis Over 6 Periods
Description: Total Tic Severity Score on the the Yale Global Tic Severity Scale - Part 2 only (lower is better), range 0 - 50
Time Frame: 3 week period of treatment
Population: All Part 2 participants
Measure: Least Squares Mean (Standard Error); unit: Total Tic Severity Score
Groups:
- AZD5213 0.5 mg: Part 1 single dose, Part 2 - multiple 3 week treatment periods in a randomized 6 period crossover design
- AZD5213 2.0 mg: Part 2 - multiple 3 week treatment periods in a randomized 6 period crossover design
- Placebo: Part 2 - multiple 3 week treatment periods in a randomized 6- period crossover design
Arm/Group | AZD5213 0.5 mg | AZD5213 2.0 mg | Placebo
Number analyzed (Participants) | 23 | 19 | 21
Total Tic Severity Score | 24.32 (2.01) | 25.41 (2.05) | 22.99 (2.03)
Statistical Analysis 1: Comparison: AZD5213 2.0 mg vs Placebo; Comparison with placebo; Test type: Superiority or Other; p = 0.0087, ANCOVA — Bonferroni-Holm adjustment, compared with 0.025; Each subject received each treatment multiple times in a crossover design; Mean Difference (Net) = 2.42, Standard Error of Mean 0.90
Statistical Analysis 2: Comparison: AZD5213 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.1198, ANCOVA — Bonferroni-Holm compared with 0.025; Each subject received each treatment multiple times in a crossover design; Median Difference (Net) = 1.34, Standard Error of Mean 0.85

2. Primary Outcome: Pharmacokinetics : Maximum Plasma Concentration (ng/ml) - Part 1 Only
Description: Pharmacokinetics Part 1 only: Maximum plasma Concentration (ng/ml) Single dose Day 1 AZD5213 0.5 mg
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: Plasma concentration (ng/ml)
Arm/Group | AZD5213 0.5 mg
Number analyzed (Participants) | 23
Plasma concentration (ng/ml) | 3.690 (1.405)

3. Primary Outcome: Pharmacokinetics : Time to Maximum Concentration (hr) - Part 1 Only
Description: Pharmacokinetics Part 1 only: Time to maximum plasma concentration (hr)Single dose Day 1 AZD5213 0.5 mg
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: Time (hr)
Arm/Group | AZD5213 0.5 mg
Number analyzed (Participants) | 23
Time (hr) | 2.112 (1.004)

4. Primary Outcome: Pharmacokinetics : AUC (h*ng/ ml) - Part 1 Only
Description: Pharmacokinetics Part 1 only: Single dose Day 1 AZD5213 0.5 mg Area Under the Concentration time curve (AUC) 0 to infinity (h*ng/ml)
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: AUC (h*ng/ml)
Arm/Group | AZD5213 0.5 mg
Number analyzed (Participants) | 23
AUC (h*ng/ml) | 26.356 (9.155)

ADVERSE EVENTS:
Time Frame: 176 days
Description: Part 1 - Single dose Day 1 - multiple dose day 6-8 Part 2 - Six period crossover Day 9 -176
Groups:
- Part 1 - AZD5213 0.5 mg: Part 1 - Day 1, AZD5213 0.5 mg
- Part 1 - AZD5213 2.0 mg: Part 1 - Days 6-8, AZD5213 2.0 mg
- Part 2 - AZD5213 0.5 mg: Part 2 - AZD5213, 0.5 mg periods (2-4 periods)
- Part 2 - AZD5213 2.0 mg: Part 2 - AZD5213, 2.0 mg periods (2 periods)
- Part 2 - Placebo: Part 2 - Placebo periods (2 periods)
- Part 1 - Placebo: Part 1 - Placebo, Days 2-5, washout after 0.5 mg single dose
Arm/Group | Overall Study | Part 1 - AZD5213 0.5 mg | Part 1 - AZD5213 2.0 mg | Part 2 - AZD5213 0.5 mg | Part 2 - AZD5213 2.0 mg | Part 2 - Placebo | Part 1 - Placebo
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/24 | 1/24 | 0/23 | 0/19 | 1/21 | 0/24
Other Adverse Events (participants affected / at risk) | 22/24 | 1/24 | 7/24 | 16/23 | 9/19 | 11/21 | 5/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Overall Study (N=24) | Part 1 - AZD5213 0.5 mg (N=24) | Part 1 - AZD5213 2.0 mg (N=24) | Part 2 - AZD5213 0.5 mg (N=23) | Part 2 - AZD5213 2.0 mg (N=19) | Part 2 - Placebo (N=21) | Part 1 - Placebo (N=24)
Testicular torsion (Part 2) (Reproductive system and breast disorders) | 1/23 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Surgical orchiectomy required, treatment continued (placebo treatment period)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Overall Study (N=24) | Part 1 - AZD5213 0.5 mg (N=24) | Part 1 - AZD5213 2.0 mg (N=24) | Part 2 - AZD5213 0.5 mg (N=23) | Part 2 - AZD5213 2.0 mg (N=19) | Part 2 - Placebo (N=21) | Part 1 - Placebo (N=24)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tic (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Abnormal behavior (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impulsive behavior (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervigilance (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sexually inappropriate behavior (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (17) | 0 (0) | 2 (2) | 5 (8) | 2 (3) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 3 (5) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (8) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Feeling abnormal (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orapharangeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0/18 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (10) | 1 (1) | 3 (3) | 1 (4) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days